CLINICAL TRIAL: NCT06578442
Title: Determining the Effect of Electromagnetic Field Treatment on Individuals With Chronic Constipation: Randomized Controlled Study
Brief Title: Effectiveness of Electromagnetic Field Therapy in Chronic Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Dilanur Özkaraoğlu, PT, MSc, Assistant Professor, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MedipolU-FTR-DO-03
Record Dates: First submitted 2024-03-12; First posted 2024-08-29 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Constipation; Electrotherapy
Keywords: Quality of Life; Magnetic Fields
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: Two groups with a conventional therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Magnetic Field Treatment was applied to the participants for 30 minutes a day, twice a week for 8 weeks, using an electromagnetic field therapy device, in a supine position, by placing circular magnetotherapy electrodes in the abdominal area, at 25 Hz and 30 Gauss power.
  Interventions: Other: Magnetic Field Treatment
- Control group (Experimental): The control group was given "constipation coping training" and asked to perform the taught methods every day for 8 weeks. Whether the individuals applied the methods was checked every day via telerehabilitation.
  Interventions: Other: Constipation Coping Training

INTERVENTIONS:
Other: Magnetic Field Treatment — Magnetic Field Treatment was applied to the participants for 30 minutes a day, twice a week for 8 weeks, using an electromagnetic field therapy device, in a supine position, by placing circular magnetotherapy electrodes in the abdominal area, at 25 Hz and 30 Gauss power.
  Arms: Treatment group
Other: Constipation Coping Training — The control group was given "constipation coping training" and asked to perform the taught methods every day for 8 weeks. Whether the individuals applied the methods was checked every day via telerehabilitation.
  Arms: Control group

SUMMARY:
The aim of the study is to examine the effects of magnetic field therapy on individuals with chronic constipation. 40 individuals with chronic constipation between the ages of 18-68 who met the inclusion criteria were included in the study. Participants were divided into two groups: treatment group (n=20) and control group (n=2O). The control group was given "constipation coping training" and asked to perform the taught methods every day for 8 weeks. Whether the individuals applied the methods was checked via telehabilitation. Participants in the treatment group received magnetic field therapy twice a week for 8 weeks. Participants were evaluated with the Constipation Severity Scale, Constipation Quality of Life Scale and International Physical Activity Questionnaire before and after the treatment.

Magnetic field therapy provides improvement in sub-parameters such as difficulty in defecation, slowing down of colon movements, and pain due to constipation. It has provided an increase in the quality of life due to constipation. Magnetic field therapy can be applied as an alternative treatment method for the treatment of individuals with chronic constipation problems.

DETAILED DESCRIPTION:
This study was carried out in the laboratory of Istanbul Medipol University Physiotherapy and Rehabilitation department on participants between February 2019 and January 2020 and were diagnosed with chronic constipation.

This study was conducted in accordance with the principles of human experimentation specified in the Declaration of Helsinki and with ethics committee approval. Informed consent forms were obtained from the participants.

52 participants were included in our study. The study was completed with 40 participants. Evaluations were made twice, before and after treatment. Magnetic field treatmentwas applied to the participants for 30 minutes a day, twice a week, for 8 weeks, using an electromagnetic field therapy device, in a supine position, by placing circular magnetic field treatment electrodes in the abdominal area, at a power of 25 Hz and 30 Gauss. Participants were informed about the things to consider in magnetic field treatment. To determine the effectiveness of the treatment, evaluations were made before and after the treatment using the Constipation Severity Scale, Constipation Quality of Life Scale, International Physical Activity Questionnaire.

Magnetic field therapy provided improvement in subparameters such as difficulty in defecation, slowing of colon movements, pain due to constipation and increased quality of life due to constipation.

ELIGIBILITY:
Inclusion Criteria:

* Presence of chronic constipation according to Rome III criteria
* Ages of 18-68
* Indicate magnetotherapy treatment,
* Not having used any medication for constipation during the treatment
* Fully cooperative

Exclusion Criteria:

* Severely obese patients
* Electrical implants in their body
* First trimester of pregnancy
* Implanted inner ear implants
* Small implants that may be affected by the magnetic field
* Epilepsy
* Untreated hypertoid
* High fever

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Constipation Severity Scale (CSS) | Four weeks
  It is a scale that reveals the symptoms of constipation in people. It makes an evaluation to determine the problems experienced by individuals in defecation. The scale includes 16 questions. The lowest total score that can be obtained from the scale is 0 and the highest is 73. A high score indicates that the symptoms are serious.
Constipation Quality of Life Scale | Four weeks
  It is a self-rating scale consisting of worry/anxiety, physical discomfort, psychosocial discomfort and satisfaction subscales. Item scores of the Likert-type scale vary between 1-5. The highest score that can be obtained from the scale is 140 and the lowest score is 28. A high score indicates poor quality of life.

SECONDARY OUTCOMES:
International Physical Activity Survey-Short Form (IPAQ-SF) | Four weeks
  Physical activities performed for at least 10 minutes at a time are evaluated. Made in the last 7 days; Vigorous physical activities and their duration (football, basketball, aerobics, fast cycling, etc.), moderate physical activities and their duration (light load carrying, cycling at normal speed, folk dances, etc.), walking and one-day sitting times are questioned and noted. All activities performed are converted to MET and the total physical activity score (MET×min×week) is calculated. According to the total physical activity score, participants' physical activity levels are classified as "low, medium and high".

CONTACTS AND LOCATIONS:
Overall Officials: Esra Atilgan, PhD, Principal Investigator — Medipol University; Gizem Boztas Elverisli, PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No